CLINICAL TRIAL: NCT04150679
Title: Hepaticojejunostomy With or Without Permanent Duodenal Access Loop in Treatment of Iatrogenic Bile Ducts Injuries, a Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hazem Nour Abdellatif, Assistant professor, Zagazig University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Hazem Nour access loop
Record Dates: First submitted 2019-10-31; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-10

CONDITIONS: Iatrogenic Bile Duct Injuries; Duodenojejunostomy Access Loop
Keywords: bile duct injury; duodenal access; hepaticojejonostomy

STUDY DESIGN:
Intervention Model Description: group I, retrospective group , data retrieved from medical records, cases treated with hepaticojejunostomy without access group II prospective group cases treated with hepaticojejunostomy with access
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group I retrospective non access loop (Active Comparator): patients with iatrogenic bile duct injuries, cases treated with hepaticojejunostomy without access loop
  Interventions: Procedure: hepaticojejunostomy without access loop
- GROUP II access loop group (Active Comparator): patients with iatrogenic bile duct injuries, cases treated with hepaticojejunostomy with duodenojejunostomy access loop
  Interventions: Procedure: duodenojejunostomy access loop

INTERVENTIONS:
Procedure: duodenojejunostomy access loop — ROUX en Y hepaticojejunostomy with duodenojejunal anastomosis as permanent access
  Arms: GROUP II access loop group
Procedure: hepaticojejunostomy without access loop — ROUX en Y hepaticojejunostomy without access loop
  Arms: group I retrospective non access loop

SUMMARY:
A comparative study between two groups, group I; retrospective group, 21 patients underwent hepaticojejunostomy for treatment of iatrogenic bile duct injuries without access loop, in the period between January 2013 and December 2014, group II; a prospective group, 23 patients underwent hepaticojejunostomy for iatrogenic bile duct injuries with duodenojejunostomy as a permanent access loop, in the period between June 2017 and May 2019. Primary (early and late outcome) and management of complications data were collected and analyzed properly.

DETAILED DESCRIPTION:
This study is a comparative study, comparing between two groups of patients with post cholecystectomy biliary injury, group (I) 21 patients, a retrospective group where data was collected from the medical records of the patients presented with post cholecystectomy biliary injury and managed with hepaticojejunostomy without access loop in a period of 2 years between January 2013 and December 2014, and group (II) 23 patients, a prospective group, where patients presented with post cholecystectomy biliary injury in a 2 years period between January 2017 and December 2018 , and managed by hepaticojejunostomy and jejunoduodenostomy as a permanent access loop .

the data collected from both groups included, demographic criteria of patients, type of the previous surgery, place of surgery, the class of the biliary injury according to bismuth classification, (according to Bismuth classification; type I (Low injury, stump length > 2 cm), type II) (higher injury, stump length < 2 cm), type III (high CHD injury but confluence is preserved), type IV (high injury both hepatic ducts are no more connected.). And any diagnostic or therapeutic intervention carried out before surgical management.

The detailed surgical management; in group I a roux en y hepaticojejunostomy was done, after abdominal exploration and identification of the level of injury or stricture a ROUX en Y loop of the jejunum was prepared 40 cm post duodenojujenal junction, it was separated and anastomosed to the jejunum at a more distal point ( 60 cm ) the proximal end of the distal loop was closed in two layers with Vicryl 3\0 the loop was extracted retrocolic towards the site of injury where a hepaticojejunostomy was done end( biliary)to side (jejunum with Vicryl 4\0 size single layer .

in the second group the same was done but with jejunoduodenostomy side to side at 5-10 cm distal to the site of hepaticoduodenostomy as a permanent access loop.

Follow up data either clinical, laboratory or radiologic were collected, findings of MRCP (if needed) was reported as primary outcome.

Secondary outcome (management of complications), including the operative time needed for correction of the complications, early and late postoperative morbidity and mortality.

The data was analyzed properly using SPSS 18, and presented in a suitable way using graphs figures and tables.

ELIGIBILITY:
Inclusion Criteria:

• Iatrogenic bile duct injuries

Exclusion Criteria:

• Hepatobiliary malignancies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
results management of biliary enteric anastomosis complications | 2 years
  access loop used as a way for endoscopic management of complications

SECONDARY OUTCOMES:
postoperative complications | ( 1st month post operative)
  Peritoneal collection Bile leak Wound infection Biliary stricture Recurrent cholangitis 2ry biliary cirrhosis Incisional hernia

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig Faculty of Medicine, Zagazig, Sharqya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided